CLINICAL TRIAL: NCT07003568
Title: Practical Clinical Study of Dual-targeting BCMA-GPRC5D CAR-T Cell Therapy for Extramedullary Infiltration in Refractory/Relapsed Multiple Myeloma
Brief Title: Dual-target BCMA-GPRC5D CAR-T Cell Therapy for RR/MM With Extramedullary Infiltration
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Collaborators: Shanghai Liquan Hospital (Other); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jing Pan, Director of the department of Immunotherapy for Hematopoietic Malignancies, Beijing GoBroad Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJGBYY-IIT-LCYJ-2025-030
Record Dates: First submitted 2025-05-23; First posted 2025-06-04 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Relapsed or Refractory Multiple Myeloma (RRMM)
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dual-targeting BCMA-GPRC5D CAR-T cell therapy (Experimental): Patients receive dual-targeting BCMA-GPRC5D CAR-T cell therapy
  Interventions: Drug: Dual-targeting BCMA-GPRC5D CAR-T cell infusion

INTERVENTIONS:
Drug: Dual-targeting BCMA-GPRC5D CAR-T cell infusion — Approximately 3-5 days prior to BCMA-GPRC5D CAR-T cell infusion, subjects are treated with FC regimen (fludarabine and cyclophosphamide) for lymphodepletion. CAR-T cell infusion are performed 48 h after completion of chemotherapy.

SUMMARY:
This is a multicenter, open-label, non-randomized, single-arm clinical trial. Patients with relapsed/refractory multiple myeloma accompanied by extramedullary infiltration will receive BCMA - GPRC5D CAR-T cell therapy.

The primary objective is to prospectively evaluate the safety of dual-targeting BCMA and GPRC5D CAR - T cell therapy for extramedullary infiltration in relapsed/refractory multiple myeloma. The primary endpoints are to assess the type and incidence of dose-limiting toxicity (DLT) within one month after the reinfusion of BCMA-GPRC5D CAR-T cells in patients, as well as the incidence and severity of adverse events within one month after the reinfusion. It is expected that no more than 18 participants will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the trial and have good compliance.
2. Aged between 18 and 75 years old, regardless of gender.
3. Diagnosed with relapsed or refractory multiple myeloma according to the criteria of the International Myeloma Working Group (IMWG)2, and have measurable extramedullary lesions due to multiple myeloma.
4. Positive for BCMA and GPRC5D in flow cytometry of bone marrow or cerebrospinal fluid tumor cells or immunohistochemistry of tumor tissue.
5. Organ functions: ① Cardiac function: Left ventricular ejection fraction > 50% (by echocardiogram) in the past 2 weeks. ② Liver function: Alanine aminotransferase and aspartate aminotransferase < 3 times the upper limit of normal (ULN). ③ Renal function: Creatinine clearance rate ≥ 40 mL/min (by Cockcroft and Gault formula). ④ Coagulation function: PT and APPT < 1.5 times the ULN. ⑤ Arterial oxygen saturation (SpO₂) > 95%. ⑥ Pulmonary function: FEV₁% predicted value ≥ 50%.
6. Female patients of childbearing age must have a negative serum pregnancy test at screening and before receiving cyclophosphamide and fludarabine or melphalan treatment; male patients should be willing to use effective contraceptive methods for 1 year after receiving the study treatment.
7. ECOG score ≤ 2.
8. Expected survival time > 3 months.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Active infections that have not been effectively controlled.
3. Active autoimmune diseases that have not been effectively controlled.
4. Adverse reactions caused by previous treatments have not recovered to CTCAE grade ≤ 1.
5. For allogeneic transplant patients, active graft - versus - host disease (GVHD) that has not been effectively controlled.
6. Presence of any of the following: HBV - DNA copy number above the lower limit of detection; positive hepatitis C antibody (HCV - Ab) with HCV - RNA copy number above the lower limit of measurability; positive anti - Treponema pallidum antibody (TP - Ab); positive human immunodeficiency virus (HIV) antibody test.
7. Allergic or intolerant to fludarabine or cyclophosphamide.
8. Suffering from known symptomatic non - plasma cell infiltrative central nervous system diseases.
9. Uncontrollable cardiovascular and cerebrovascular diseases within 6 months, such as: a. New York Heart Association (NYHA) class III or IV congestive heart failure. b. Myocardial infarction occurred or coronary artery bypass grafting (CABG) was received ≤ 6 months before enrollment. c. Clinically significant ventricular arrhythmia or a history of unexplained syncope (excluding cases caused by vasovagal or dehydration). d. A history of severe non - ischemic cardiomyopathy.
10. A history of other untreated malignancies within the past 5 years or having other untreated malignancies concurrently.
11. The investigator assesses that the subject cannot or is unwilling to comply with the requirements of the study protocol.
12. Previous use of a CAR - T vector with the same structure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2027-05-25 (Estimated); Study Completion 2027-06-25 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 30 days
  Incidence and type of dose-limiting toxicity(DLT) within 1 month of BCMA-GPRC5D CAR-T infusion.
Adverse events (AEs） | 30 days
  Total number, incidence and severity of adverse events (AEs) within 30 days of BCMA-GPRC5D CAR-T infusion

SECONDARY OUTCOMES:
Overall remission rate (ORR) | 90 days
  The assessment of ORR by dose group at 90 Days after BCMA-GPRC5D CAR-T infusion.
Event Free Survival (EFS) | from enrollment to the end of treatment at 2 years
  Evaluate the EFS of dual-targeting BCMA-GPRC5D CAR-T cell therapy for extramedullary infiltration in relapsed and refractory multiple myeloma
Duration of Response (DOR) | from enrollment to the end of treatment at 2 years
  Evaluate the DOR of dual-targeting BCMA-GPRC5D CAR-T cell therapy for extramedullary infiltration in relapsed and refractory multiple myeloma
Overall Survival (OS) | from enrollment to the end of treatment at 2 years
  Evaluate the OS of dual-targeting BCMA-GPRC5D CAR-T cell therapy for extramedullary infiltration in relapsed and refractory multiple myeloma

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Liquan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided